CLINICAL TRIAL: NCT06810921
Title: Lateral Sinus Augmentation Utilizing Bovine Bone Mixed with Platelet-rich Fibrin: Evaluation of Graft Volume Changes Based on CBCT Imaging
Brief Title: Lateral Sinus Augmentation Utilizing Bovine Bone Mixed with Platelet-rich Fibrin
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, NIBRAS HAMDAN CHASIB BAIDHANI, lecturer at University of Baghdad, University of Baghdad
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 998125
Record Dates: First submitted 2025-01-27; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Lateral Sinus Lifting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- utilizing bovine bone mixed with PRF for sinus lifting (Active Comparator)
  Interventions: Procedure: lateral sinus lift

INTERVENTIONS:
Procedure: lateral sinus lift — A rectangular shaped osteotomy was performed using a low-speed surgical handpiece and round diamond bur, with copious cooled normal saline irrigation.
  The Schneiderian membrane (SM) was gently elevatated using Frios Sinus Set elevators for implant placement

SUMMARY:
Background:

In sinus augmentation procedure, graft resorption remains a major dilemma of various graft materials.

Objective:

To estimate the graft volume changes following lateral sinus augmentation utilizing cone beam computed tomography.

Methods: A total of 34 lateral sinus augmentation operations were performed and 50 dental implants were concomitantly inserted. The sinus augmentation cases were distributed randomly into 3 groups according to graft material: Group A comprised utilizing deproteinized bovine bone alone, group B using deproteinized bovine bone mixed with leukocyte and platelet-rich fibrin, and group C employing deproteinized bovine bone mixed with advanced platelet-rich fibrin. Cone-beam computed tomography was obtained 2 weeks (baseline record) and 24 weeks postoperatively for the measurement of the graft volume changes.

ELIGIBILITY:
Inclusion Criteria:

* requiring lateral sinus lift for implant placement

Exclusion Criteria:

* available bone permits implant placement without need for sinus lifting

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of graft volume changes based on CBCT imaging | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, Bab Al Muadham, Baghdad Governorate, Iraq

IPD SHARING:
Plan to Share IPD: Undecided